CLINICAL TRIAL: NCT05891249
Title: A Phase 4 Study to Evaluate Safety and Effectiveness of Luspatercept (ACE-536) for the Treatment of Anemia Due to IPSS-R Very Low, Low, or Intermediate Risk Myelodysplastic Syndromes (MDS) With Ring Sideroblasts Who Require Red Blood Cell Transfusions in Participants Who Have Had Unsatisfactory Response to or Are Ineligible to Erythropoietin Based Therapy and in Participants With Transfusion Dependent Anemia Due to Beta-Thalassemia
Brief Title: A Study to Evaluate the Safety and Effectiveness of Luspatercept for the Treatment of Transfusion-dependent (TD) Anemia Associated With Myelodysplastic Syndromes (MDS) & Beta-thalassemia (β-Thal) in India
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA056-023
Record Dates: First submitted 2023-05-26; First posted 2023-06-06 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Anemia
Keywords: Luspatercept; ACE-536; Transfusion dependent; Beta-thalassemia; Myelodysplastic syndromes with ring sideroblasts; Anemia; Hemoglobinopathies; Hematologic diseases; Bone marrow diseases
MeSH Terms: conditions — Anemia; beta-Thalassemia; Hemoglobinopathies; Hematologic Diseases; Bone Marrow Diseases | interventions — luspatercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Luspatercept (Experimental)
  Interventions: Biological: Luspatercept

INTERVENTIONS:
Biological: Luspatercept — Specified dose on specified days
  Other Names: ACE-536; REBLOZYL; BMS-986346; ROJUZDA

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of luspatercept in participants who require regular blood cell transfusions due to b-thalassemia and myelodysplastic syndromes in India

ELIGIBILITY:
Inclusion Criteria:

β-Thalassemia Cohort

* Documented diagnosis of β-thalassemia or hemoglobin (Hb E/β-thalassemia). (β-thalassemia with mutation and/or multiplication of alpha [α] globin is allowed).
* Regularly transfused, defined as 6 RBC units to 20 RBC units in the 24 weeks prior to enrollment and no transfusion-free period for > 35 days during that period.

MDS-RS Cohort

- Participant has documented diagnosis of MDS according to World Health Organization (WHO) (2016)/French-American-British FAB classification that meets revised International Prognostic Scoring System (IPSS-R) classification of very low, low, or intermediate risk disease and the following criteria: i) RS ≥ 15% of erythroid precursors in bone marrow. If the SF3B1 mutation is present, RS ≥ 5% will be included.

ii) Less than 5% blasts in bone marrow and < 1% peripheral blood blasts. iii) Peripheral blood white blood cell (WBC) count < 13,000/ microliters (μL).

* If the participant was previously treated with erythropoiesis-stimulating agents (ESAs) or granulocyte colony-stimulating factor (G-CSF)/granulocyte-macrophage colony-stimulating factor (GM-CSF), both agents must have been discontinued ≥ 4 weeks prior to the date of enrollment.

Exclusion Criteria:

β-Thalassemia Cohort

* A diagnosis of Hb S/β-thalassemia or α-thalassemia (for exampe, Hemoglobin H).
* Deep vein thrombosis (DVT) or stroke requiring medical intervention ≤ 24 weeks prior to enrollment.
* Use of chronic anticoagulant therapy is excluded unless the treatment stopped at least 28 days prior to enrollment. Anticoagulant therapies used for prophylaxis for surgery or high-risk procedures as well as low-molecular-weight (LMW) heparin for superficial venous thrombosis and chronic aspirin are allowed.
* Cytotoxic agents or immunosuppressants or immunomodulatory drugs (IMiDs) ≤ 28 days prior to enrollment (ie, antithymocite globulin or cyclosporine or thalidomide).

MDS-RS Cohort

* MDS associated with del 5q cytogenetic abnormality.
* Secondary MDS, that is, MDS that is known to have arisen as the result of chemical injury or treatment with chemotherapy and/or radiation for other diseases.
* Participant has known clinically significant anemia due to iron, vitamin B12, or folate deficiencies; autoimmune or hereditary hemolytic anemia; or gastrointestinal bleeding.
* Iron deficiency to be determined by serum ferritin ≤ 15 micrograms per liter (μg/L) and additional testing if clinically indicated (for example, calculated transferrin saturation [iron/total iron binding capacity ≤ 20%] or bone marrow aspirate [BMA] stain for iron).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2023-06-05 (Actual); Primary Completion 2028-12-16 (Estimated); Study Completion 2028-12-16 (Estimated)

PRIMARY OUTCOMES:
β-Thal Cohort: Number of participants with treatment-related adverse events (AEs) of grade 3 or higher | Up to 57 weeks
MDS-Ring Sideroblasts (RS) Cohort: Number of participants with treatment-related AEs of grade 3 or higher | Up to 54 weeks

SECONDARY OUTCOMES:
β-Thal Cohort: Percentage of participants who achieved red blood cell (RBC) transfusion burden reduction (≥ 33% reduction from baseline) with a reduction of at least 2 red cell units compared to the 12-week interval prior to enrollment | Week 13 to week 24
β-Thal Cohort: Percentage of participants who achieved RBC transfusion burden reduction of at least 33% from baseline during any 12-week interval with a reduction of at least 2 red cell units compared to the 12-week interval prior to enrollment | Up to 57 weeks
MDS-RS Cohort: Percentage of participants who achieved RBC-TI during any consecutive 56-day period | Week 1 to week 24
β-Thal Cohort: Number of participants with treatment-related AEs | Up to 57 weeks
MDS-RS Cohort: Number of participants with treatment-related AEs | Up to 54 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (9):
- India (9):
  - Local Institution - 0002, Ahmedabad, Gujarat
  - Local Institution - 0001, New Delhi, National Capital Territory of Delhi
  - Local Institution - 0007, Kolkata, West Bengal
  - Local Institution - 0005, Assam
  - Local Institution - 0003, Bangalore
  - Local Institution - 0004, Chandigarh
  - Local Institution - 0010, Delhi
  - Local Institution - 0006, Hyderabad
  - Local Institution - 0008, Mumbai

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html